CLINICAL TRIAL: NCT01231321
Title: An Open-label, Prospective, Multi-Centre Study to Assess the Safety and Efficacy of Adalimumab (Humira®) When Added to Inadequate Standard Anti-Rheumatic Therapy in Patients With Active Rheumatoid Arthritis
Brief Title: A Study of Adalimumab When Added to Inadequate Standard Anti-rheumatic Therapy in Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Konstantin Gudkov/ Clinical Research Manager, Abbott Laboratories LLC Russia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W06-406
Record Dates: First submitted 2010-10-28; First posted 2010-11-01 (Estimated); Results first posted 2011-03-24 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Adalimumab added to inadequate standard anti-rheumatic therapy in patients with active Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- adalimumab (Experimental): Adalimumab / pre-filled syringe 40 mg/0.8 ml
  Interventions: Drug: adalimumab

INTERVENTIONS:
Drug: adalimumab — Adalimumab 40 mg in 0.8 ml in pre-filled syringe for under the skin of the abdomen or the thigh injection every other week.
  Other Names: ABT-D2E7; Humira

SUMMARY:
A total of 100 participants diagnosed with active rheumatoid arthritis were enrolled at 5 sites in Russia. Adalimumab was administered by subcutaneous injection every other week, with dose escalation to weekly dosing available for participants not receiving concomitant disease-modifying antirheumatic drugs (DMARDs) who did not achieve American College of Rheumatology 20 (ACR20) criteria after 12 weeks of treatment. Efficacy and safety measurements were performed throughout the study.

DETAILED DESCRIPTION:
This is an open-label, multicenter study designed to establish the safety and efficacy of adalimumab in the treatment of moderate to severely active rheumatoid arthritis. A total of 100 subjects with inadequate preexisting standard anti-rheumatic therapy were enrolled at 5 sites in Russia.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females >= 18 years of age.
2. A negative pregnancy test (human chorionic gonadotropin in serum samples) for women of childbearing potential prior to start of study treatment.
3. Female subject is either not of childbearing potential, defined as postmenopausal (at least 1 year since last menses) or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or is of childbearing potential and practicing one of the following methods of birth control throughout the study and for 150 days after study completion:

   * Condoms, sponge, foams, jellies, diaphragm or intrauterine device.
   * Contraceptives (oral, parenteral, patch) for three months prior to study drug administration.
   * A vasectomized partner.
4. American College of Rheumatology criteria for diagnosis of rheumatoid arthritis for at least 6 months.
5. Subjects must meet the following three criteria:

   * Disease Activity Score (28 joints) more or equal 3.2 (at Baseline only)
   * At least 6 swollen joints out of the 66 assessed
   * At least 8 tender joints out of the 68 assessed
6. Subjects must have a C-reactive protein >= 1.5mg/dL or erythrocyte sedimentation rate >= 28 mm/1h.
7. Unsatisfactory response or intolerance to prior disease modifying anti-rheumatic drugs (must have failed at least 1 disease modifying anti-rheumatic drug).
8. Able and willing to administer subcutaneous injections.
9. Able and willing to give written informed consent and to comply with the requirements of the study protocol.
10. Documented negative purified protein derivative test, defined as < 5 mm induration, or willingness and ability to start tuberculosis prophylaxis before first dose of study drug if the purified protein derivative result is positive and the chest X-ray is not suggestive of active tuberculosis and there is no history of active tuberculosis.

Exclusion Criteria:

1. Prior treatment with alkylating agents such as cyclophosphamide or chlorambucil within at least 5 years before enrollment.
2. Prior treatment with intravenous immunoglobulin or any investigational agent "chemical" in nature within 30 days, or 5 half lives of the product, whichever is longer.
3. Prior treatment with cyclosporine within the last 6 months.
4. Prior treatment with investigational biologic therapy.
5. Subject has chronic arthritis diagnosis before the age 17 years.
6. Subject has undergone joint surgery within the preceding two months (at joints to be assessed within the study).
7. History of an allergic reaction or significant sensitivity to the constituents of study drug (adalimumab).
8. Treatment within the last 2 months with approved biologic therapy (e.g. infliximab) prior to Baseline.
9. Prior treatment with total lymphoid irradiation.
10. History of cancer or lymphoproliferative disease other than a successfully and completely treated non-metastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix.
11. History of or current acute inflammatory joint disease of origin other than rheumatoid arthritis, e.g. mixed connective tissue disease, systemic lupus erythematosus etc.
12. History of uncontrolled diabetes, unstable ischemic heart disease, congestive heart failure (New York Heart Association III-IV), active peptic ulcer disease, recent stroke (within 3 months) and any other condition which, in the opinion of the investigator, would put the subject at risk by participation in the protocol.
13. Subject is known to have immune deficiency, history of positive human immunodeficiency virus status or is immunocompromised.
14. Persistent chronic infection, or severe infections requiring hospitalization or treatment with intravenous antibiotics within 30 days, or oral antibiotics within 14 days prior to enrollment.
15. Female subjects who are pregnant or breast-feeding or is considering becoming pregnant during the study or for 150 days after the last dose of study medication.
16. History of clinically significant drug or alcohol abuse in the last year.
17. Previous diagnosis or signs of central nervous system demyelinating diseases.
18. History of untreated or active tuberculosis, histoplasmosis or listeriosis.
19. History of clinically significant hematologic (e.g. severe anemia, leucopenia, thrombocytopenia), renal or liver disease (e.g. fibrosis, cirrhosis, hepatitis).
20. Screening clinical laboratory analysis showing any of the following abnormal laboratory results:

    * Aspartate transaminase or alanine transaminase > 1.75 x the upper limit of normal.
    * Serum total bilirubin >= 1.5 mg/dL (>= 26 micromol/L).
    * Creatinine > 1.5 mg/dL (133 micromol/L) in subjects < 65 years old and > upper limit of normal range in subjects >= 65 years old.
    * Positive Hepatitis B or C serology indicative of previous or current infections.
21. Subject is considered by the Investigator, for any reason, to be an unsuitable candidate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin Gudkov, MD, Study Director — Abbott
Locations (5):
- Russia (5):
  - Site Ref # / Investigator 17682, Kazan'
  - Site Ref # / Investigator 7417, Moscow
  - Site Ref # / Investigator 17681, Moscow
  - Site Ref # / Investigator 7401, Moscow
  - Site Ref # / Investigator 18081, Saint Petersburg

RESULTS

PARTICIPANT FLOW:
Groups:
- Adalimumab/ Pre-filled Syringe 40 mg/0.8 mL: Adalimumab 40 mg in 0.8 ml in pre-filled syringe for under the skin of the abdomen or the thigh injection every other week.
Period: Overall Study
Arm/Group | Adalimumab/ Pre-filled Syringe 40 mg/0.8 mL
Started | 100
Completed | 95
Not Completed | 5
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Adalimumab/ Pre-filled Syringe 40 mg/0.8 mL
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 90
  >=65 years | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 50.9 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89
  Male | 11
Region of Enrollment [Number; unit: participants]
  Russian Federation | 100

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Adverse Events
Description: Serious adverse events were collected from the time of informed consent, and nonserious adverse events were collected from the time of first dose of adalimumab, until 70 days after the last injection of adalimumab. Refer to the Reported Adverse Events section of this results disclosure for specific adverse events reported.
  Note:
  Severe events considerably interfered in patients' usual activities and may have been life-threatening.
  Serious events were life-threatening; resulted in hospitalization, congenital anomalies, or disability; or required intervention to prevent seriousness.
Time Frame: Up to 34 weeks (24 week study treatment plus 70-day follow-up period)
Population: All enrolled subjects were included in this intent-to-treat (ITT) analysis.
Measure: Number; unit: participants
Arm/Group | Adalimumab/ Pre-filled Syringe 40 mg/0.8 mL
Number analyzed (Participants) | 100
participants
  Adverse events | 38
  Serious adverse events | 1
  Severe adverse events | 1
  Possibly or probably related to adalimumab | 24
  Adverse events leading to discontinuation | 3
  Fatal adverse events | 0

2. Primary Outcome: Changes of Physical Examination
Description: Physical examination findings were compared between Baseline and Week 24, and changes were recorded (Normal at Baseline to Abnormal at Week 24; or Abnormal at Baseline to Normal at Week 24). Physical examination criteria (normal vs. abnormal) were at the clinical judgement of the examining physician. Significant changes in physical examination from Baseline were considered to be adverse events.
Time Frame: Baseline and 24 weeks
Population: All enrolled subjects with available data were included in this intent-to-treat (ITT) analysis.
Measure: Number; unit: participants
Groups:
- Change From Normal to Abnormal: Subjects whose physical examination findings for the categories below were normal at Baseline and abnormal at 24 weeks
- Change From Abnormal to Normal: Subjects whose physical examination findings for the categories below were abnormal at Baseline and normal at 24 weeks
Arm/Group | Change From Normal to Abnormal | Change From Abnormal to Normal
Number analyzed (Participants) | 99 | 99
participants
  General Appearance | 0 | 0
  Head | 0 | 0
  Ears | 0 | 0
  Eyes | 1 | 0
  Nose | 0 | 0
  Throat | 0 | 0
  Neck | 0 | 0
  Thyroid | 0 | 0
  Lungs/Chest | 0 | 0
  Cardiovascular | 1 | 0
  Abdomen | 0 | 0
  Musculoskeletal | 0 | 0
  Extremities | 0 | 0
  Skin | 0 | 1
  Lymph nodes | 1 | 1
  Neurological | 0 | 0
  Genitourinary | 0 | 0
  Other | 0 | 0

3. Primary Outcome: Deviation From Normal Laboratory Ranges
Description: Laboratory values were assessed for values above and below the normal (reference) ranges used by the central laboratory.
  Note abbreviations used in table:
  Alk. phosphatase = alkaline phosphatase, ALT = alanine aminotransferase, AST = aspartate aminotransferase, ESR = erythrocyte sedimentation rate
Time Frame: 24 weeks
Population: All subjects with available data were included in this intent-to-treat (ITT) analysis. The number of subjects with available data is indicated for each laboratory assessment.
Measure: Number; unit: participants
Groups:
- Below Reference Range: Subjects with laboratory values at Week 24 lower than the reference range indicated for each parameter
- Above Reference Range: Subjects with laboratory values at Week 24 higher than the reference range indicated for each parameter
Arm/Group | Below Reference Range | Above Reference Range
Number analyzed (Participants) | 100 | 100
participants
  Basophils (%) (ref. range: 0% - 1%) (n = 95) | 0 | 0
  Basophils (ref. range 0 - 2 x 10^9/L) (n = 94) | 0 | 0
  Eosinophils (%) (ref. range 1% - 5%) (n = 95) | 17 | 11
  Eosinophils (ref. range 0 - 1 x 10^9/L) (n = 94) | 0 | 0
  Erythrocytes (ref. range 4 - 5 x 10^12/L) (n = 95) | 15 | 9
  ESR (ref. range 0 - 30 mm/h) (n = 75) | 0 | 14
  Hematocrit (ref. range 35% - 47%) (n = 95) | 15 | 2
  Hemoglobin (ref. range 12 - 16 g/dL) (n = 95) | 33 | 1
  Leucocytes (ref. range 4 - 11 x 10^3/L) (n = 95) | 3 | 10
  Lymphocytes (%) (ref. range 19% - 37%) (n = 95) | 15 | 24
  Lymphocytes (ref. range 2 - 4 x 10^9/L) (n = 94) | 44 | 6
  Monocytes (%) (ref. range 3% - 11%) (n = 95) | 1 | 12
  Monocytes (ref. range 0 - 1 x 10^9/L) (n = 94) | 0 | 6
  Neutrophils (%) (ref. range 48% - 78%) (n = 95) | 20 | 6
  Neutrophils (ref. range 2 - 9 x 10^9/L) (n = 95) | 5 | 3
  Platelets (ref. range 150-400 x 10^3/mcL) (n = 95) | 0 | 9
  Albumin (ref. range 35 - 50 g/L) (n = 97) | 0 | 14
  Alk. phosphatase (ref. range 40-150 U/L) (n = 97) | 1 | 2
  ALT (ref. range 0 - 31 U/L) (n = 97) | 0 | 9
  AST (ref. range 0 - 31 U/L) (n = 97) | 0 | 6
  Calcium (ref. range 2 - 3 mmol/L) (n = 97) | 1 | 0
  Chloride (ref. range 98 - 107 mEq/L) (n = 96) | 0 | 0
  Creatine kinase (ref. range 0 - 167 U/L) (n = 97) | 0 | 2
  Creatinine (ref. range 53 - 97 mcmol/L) (n = 97) | 1 | 1
  C-reactive protein (ref. range 0-5 mg/L) (n = 97) | 0 | 45
  Glucose (ref. range 4- 6 mmol/L) (n = 97) | 4 | 10
  Potassium (ref. range 4 - 6 mmol/L) (n = 97) | 21 | 0
  Sodium (ref. range 136 - 145 mmol/L) (n = 97) | 2 | 0
  Total bilirubin (ref. range 3-20 mcmol/L) (n = 97) | 0 | 5
  Total cholesterol (ref. range 4-8 mmol/L) (n = 97) | 5 | 4
  Total protein (ref. range 64-83 g/L) (n = 97) | 3 | 2
  Urea (ref. range 2 - 6 mmol/L) (n = 96) | 0 | 30
  Urea nitrogen (ref. range 6 - 20 mg/dL) (n = 97) | 0 | 11
  Uric acid (ref. range 150 - 350 mcmol/L) (n = 97) | 11 | 6
  Urine pH (ref. range 5 - 8) (n = 98) | 0 | 1

4. Primary Outcome: Vital Sign Values
Description: Vital signs values were assessed for values above and below the normal (reference) ranges used by the central laboratory.
  Note, in table, BP = blood pressure.
Time Frame: 24 weeks
Population: All subjects with available data were included in this intent-to-treat (ITT) analysis.
Measure: Number; unit: participants
Groups:
- Below Reference Range: Subjects with vital sign values at Week 24 lower than the reference range indicated for each parameter
- Above Reference Range: Subjects with vital sign values at Week 24 higher than the reference range indicated for each parameter
Arm/Group | Below Reference Range | Above Reference Range
Number analyzed (Participants) | 99 | 99
participants
  Systolic BP (ref. range 100 - 140 mm Hg) | 1 | 2
  Diastolic BP (ref. range 60 - 100 mm Hg) | 0 | 0
  Pulse (ref. range 50 - 90 beats/min) | 0 | 0
  Body temperature (ref. range 36 - 37 degrees C) | 1 | 0

5. Secondary Outcome: Change in Disease Activity Score (DAS28) Compared With Baseline
Description: The DAS28 is validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, C-reactive protein, and general health (patient's global assessment of disease activity) were included in the DAS28 score. Scores on the DAS28 range from 1 (inactive disease) to 10 (very active disease).
Time Frame: Baseline and 24 weeks
Population: All subjects with data available from both Baseline and Week 24 were included in this intent-to-treat (ITT) analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab/ Pre-filled Syringe 40 mg/0.8 mL
Number analyzed (Participants) | 96
units on a scale | -2.74 (1.18)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent up to 70 days after the last injection of adalimumab.
Arm/Group | Adalimumab/ Pre-filled Syringe 40 mg/0.8 mL
Serious Adverse Events (participants affected / at risk) | 1/100
Other Adverse Events (participants affected / at risk) | 38/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab/ Pre-filled Syringe 40 mg/0.8 mL (N=100)
Pyogenic arthritis (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab/ Pre-filled Syringe 40 mg/0.8 mL (N=100)
Adverse drug reaction (General disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
Arthritis bacterial (Infections and infestations) | 1
Asthenia (General disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Body temperature increased (Investigations) | 2
Bronchitis (Infections and infestations) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Ear infection (Infections and infestations) | 1
Endometriosis (Reproductive system and breast disorders) | 1
Eosinophilia (Blood and lymphatic system disorders) | 1
Furuncle (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Headache (Nervous system disorders) | 3
Herpes zoster (Infections and infestations) | 1
Herpex simplex (Infections and infestations) | 1
Injection site erythema (General disorders) | 3
Injection site pain (General disorders) | 1
Injection site papule (General disorders) | 1
Injection site pruritus (General disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Lymphocytosis (Blood and lymphatic system disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nasopharyngitis (Infections and infestations) | 4
Neutropenia (Blood and lymphatic system disorders) | 2
Oral herpes (Infections and infestations) | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 3
Pain (General disorders) | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1
Pneumonia (Infections and infestations) | 1
Pyrexia (General disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory tract infection viral (Infections and infestations) | 3
Retinopathy (Eye disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3
Rosacea (Skin and subcutaneous tissue disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
Tracheitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Wound infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.